CLINICAL TRIAL: NCT05456438
Title: Effect of Tea Tree Oil and Coconut Oil on Nipple Crack Formation in the Early Postpartum Period
Brief Title: Effect of Tea Tree Oil and Coconut Oil on Nipple Crack Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Principal Investigator,, Hitit University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-27
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Nipple Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COCONUT OİL (Experimental): * After feeding, wash hands and apply 2 drops of oil, COCONUT OİL in the 1st intervention group to the index finger and spread on the areola and nipple,
  * Continue this application for 10 days
  Interventions: Other: İntervention 1; Other: İntervention 2
- Control group (No Intervention): They were told that no intervention would be performed, and that they should not use any application like herbal or chemical oils, creams, medications, etc. on the nipples during the first 10 days postpartum.
- TEA TREE OİL (Experimental): * After feeding, wash hands and apply 2 drops of oil, TEA TREE OİL in the 2nd intervention group, to the index finger and spread on the areola and nipple,
  * Continue this application for 10 days.
  Interventions: Other: İntervention 1; Other: İntervention 2

INTERVENTIONS:
Other: İntervention 1 — Group 1 applied coconut oil to the nipple
  Other Names: application of coconut oil and tea tree oil to the nipple.
  Arms: COCONUT OİL; TEA TREE OİL
Other: İntervention 2 — Group 2 applied tea tree oil to the nipple
  Arms: COCONUT OİL; TEA TREE OİL

SUMMARY:
The aim of the study was to determine the effect of tea tree oil and coconut oil applied to the nipples during the early postpartum period on nipple crack formation.

DETAILED DESCRIPTION:
This randomized controlled experimental research included a total of 90 women in the research sample abiding by the research criteria, with 30 each in the intervention groups (coconut oil or tea tree oil application) and 30 in the control group. Women in the intervention groups applied coconut oil or tea tree oil to the nipples on the 3rd, 7th and 10th days postpartum, while the control group did not have any intervention

ELIGIBILITY:
Inclusion Criteria:

* Mothers who volunteered for participation, h
* aged from 18-45 years,
* with new and live birth after 37 weeks,
* without flat or small nipple problems,
* without previous breast operations,
* able to apply correct breastfeeding methods and with infants with birth weight of 2500 g and above were included in the study.

Exclusion Criteria:

* Mothers who could not breastfeed,
* had stillbirth,
* who had infants with congenital anomalies preventing breastfeeding were not included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
VAS Pain score | 12 months
  It is assessed on a line with 10 cm length marked at 1 cm intervals. On the scale, 0 cm represents no pain, 5 cm is moderate levels of pain and 10 cm is unbearable pain. The scale was used to assess the severity of nipple pain perceived by mothers.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Yıldırım, Çorum, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahin E, Yildirim F, Buyukkayaci Duman N. Effect of Tea Tree Oil and Coconut Oil on Nipple Crack Formation in the Early Postpartum Period. Breastfeed Med. 2023 Mar;18(3):226-232. doi: 10.1089/bfm.2022.0260. Epub 2023 Feb 10. PMID 36763614